CLINICAL TRIAL: NCT05320016
Title: Effects of Remimazolam Combined With Remifentanil on Quality of Recovery After Ambulatory Hysteroscopic Surgery: a Prospective, Observational Study
Brief Title: Effects of Remimazolam on Quality of Recovery After Ambulatory Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-2109-708-309
Record Dates: First submitted 2022-03-30; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Day Surgery; Patient Outcome Assessment; Quality of Recovery; Remimazolam
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Remimazolam — Effects of remimazolam on quality of recovery scores after ambulatory hysteroscopic surgery
  Other Names: the translated Korean version of 15-item Quality of Recovery scale (QoR-15K)

SUMMARY:
Remimazolam is a novel ultra-short acting benzodiazepine with rapid onset of effects, short maintenance and faster recovery time. Due to its recent development, few studies have investigated the effect of remimazolam on postoperative recovery mainly focusing on physiologic endpoints, recovery time and possible adverse events. Although these parameters are crucial and need evaluation, the investigators ignore quality of recovery from participant's perspective. For this purpose, various measurment tools have been developed for psychometric evaluation of QoR score.

DETAILED DESCRIPTION:
To date, there has not been a study investigating the impact of remimazolam on quality of recovery (QoR). This study evaluates the effect of remimazolam on QoR of participants undergoing general anesthesia using remimazolam-remifentanil total intravenous anesthesia (TIVA) for hysteroscopy as day surgery basis. Herein, the investigators used the translated Korean version of the 15-item Quality of Recovery-15 (QoR-15K) questionnaire, which was previously validated in Korean surgical participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman scheduled for ambulatory gynecological surgery under general anesthesia
* American Society of Anesthesiology grade 1 or 2

Exclusion Criteria:

* Underlying diseases: liver, kidney, brain nervous system, glaucoma
* Patients with BMI greater than 30 and less than 18.5
* Patients diagnosed with sleep apnea
* Alcohol or drug dependent patients
* Patients with severe or acute respiratory failure
* Lactose intolerance
* Dextran 40 hypersensitivity
* Patients in shock or coma

Ages: 19 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult woman scheduled for ambulatory gynecological surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of recovery | 24 hours after ambulatory hysteroscopic surgery
  the translated Korean version of 15-item Quality of Recovery scale (QoR-15K)

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hwan Do, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyunggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No